CLINICAL TRIAL: NCT02436096
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TNX-102 SL Tablets Taken Daily at Bedtime in Patients With Fibromyalgia
Brief Title: A Study to Evaluate eFFIcacy and Safety of Sublingual TNX-102 SL Tablet Taken at Bedtime in Patients With fibRoMyalgia
Acronym: AFFIRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-F301
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia; Myofascial Pain Syndromes; Muscular Diseases; Musculoskeletal Diseases; Nervous System Diseases; Neuromuscular Diseases; Rheumatic Diseases
Keywords: Pain; Sleep
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes; Muscular Diseases; Musculoskeletal Diseases; Nervous System Diseases; Neuromuscular Diseases; Rheumatic Diseases; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNX-102 SL Tablet, 2.8 mg (Experimental): 1 x TNX-102 SL 2.8mg Tablet taken sublingually each day at bedtime for 12 weeks
  Interventions: Drug: TNX-102 SL Tablet, 2.8mg
- Placebo SL Tablet (Placebo Comparator): 1 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks
  Interventions: Drug: Placebo SL Tablet

INTERVENTIONS:
Drug: TNX-102 SL Tablet, 2.8mg — Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 1 for 12 weeks.
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL Tablet, 2.8 mg
Drug: Placebo SL Tablet — Patients will take 1 tablet of randomly assigned study drug sublingually each day at bedtime starting on Day 1 for 12 weeks.
  Other Names: Placebo sublingual tablets
  Arms: Placebo SL Tablet

SUMMARY:
The use of low-dose CBP dosed nightly at bedtime for FM was supported by the results of Tonix' TNX-CY-F202 Phase 2b study (also referred to as the BESTFIT Study). The TNX-CY-F202 study provided evidence that TNX-102 SL 2.8 mg dosed nightly results in beneficial effects upon pain, sleep and other FM symptomatology.

The present trial is designed to assess the safety and efficacy of TNX-102 SL 2.8 mg tablets, taken daily at bedtime over 12 weeks to treat fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Fibromyalgia (2010 ACR criteria)
* Male or female 18-75 years old
* For patients with major depressive disorders only: clinically stable, no suicidal risk and stable anti-depressant therapy
* Willing and able to withdraw specific therapies (ask PI)
* Medically acceptable form of contraception (female only)
* Signed informed consent

Exclusion Criteria:

* Arthritis, lupus and other systemic auto-immune diseases
* Regional or persistent pain that could interfere with assessment of fibromyalgia pain
* Bipolar and psychotic disorders
* Increased risk of suicide
* Significant clinical (cardiac, systemic infection, systemic corticosteroid requirement, drug/alcohol abuse) or laboratory abnormalities.
* Inability to wash-out specific medications (ask PI)
* Known hypersensitivity to cyclobenzaprine
* Others: seizure disorders, severe/untreated sleep apnea, BMI>40

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Sacramento, California
  - San Diego, California
  - Brandon, Florida
  - DeLand, Florida
  - Lakeland, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Smyrna, Georgia
  - Evansville, Indiana
  - North Dartmouth, Massachusetts
  - Ann Arbor, Michigan
  - Jackson, Mississippi
  - Williamsville, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Middleburg Heights, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Warwick, Rhode Island
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Dallas, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Started | 257 | 262
Completed | 222 | 203
Not Completed | 35 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg | Total
Number analyzed (Participants) | 257 | 262 | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.20) | 47.8 (11.16) | 47.8 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 252 | 499
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 31 | 52
  Not Hispanic or Latino | 236 | 231 | 467
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 27 | 11 | 38
  White | 221 | 242 | 463
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 257 | 262 | 519

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With ≥30% Pain Improvement
Description: The primary efficacy endpoint is the proportion of patients with a ≥30% improvement (responder criteria) from baseline to Week 12 in the weekly mean of the daily self-reported 24-hour recall average pain intensity score using an 11-point (0-10) NRS. Scores range from 0 (no pain) to 10 (worst possible pain).
Time Frame: Day 1, Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
Participants | 58 | 75

2. Secondary Outcome: Patient's Global Impression of Change (PGIC)
Description: Proportion of patients with a PGIC rating of 1 ("very much improved") or 2 ("much improved") at Week 12. The PGIC is a fibromyalgia specific validated instrument on a scale of 1 to 7, where a score of 1 indicates the highest level of improvement and a score of 7 indicates the highest level of worsening.
Time Frame: Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
Participants | 42 | 62

3. Secondary Outcome: Change From Baseline to Week 12 in the Fibromyalgia Impact Questionnaire - Revised (FIQR) Symptoms Domain Score
Description: The FIQR is a validated questionnaire. Scores on the symptoms domain range from 0 to 100 where a higher score means worse outcome.
Time Frame: Day 1, Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
units on a scale | -8.2 (1.13) | -14.1 (1.14)

4. Secondary Outcome: Change From Baseline to Week 12 in the FIQR Function Domain Score
Description: The FIQR is a validated questionnaire. Scores on the function domain range from 0 to 90 where a higher score means worse outcome.
Time Frame: Day 1, Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
units on a scale | -4.4 (1.15) | -10.3 (1.16)

5. Secondary Outcome: Patient Reported Outcomes Measurement System (PROMIS) Sleep Disturbance
Description: Change from baseline in the PROMIS score for sleep disturbance at Week 12. The PROMIS Sleep disturbance short form 8a consists of 8 questions on a 5-point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40. Raw scores are converted to T-scores based on US population with score of 50 as average with a standard deviation of 10. Lower T-scores indicate less sleep disturbance.
Time Frame: Day 1, Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
T-score | -4.7 (.53) | -8.0 (.54)

6. Secondary Outcome: Weekly Average of Daily Sleep Quality Diary
Description: Change from Baseline in the weekly average of the daily diary assessment of sleep quality at Week 12. Patients provide a daily numeric assessment of their sleep quality for the previous night, via an electronic diary, using an 11-point NRS. Scores range from 0 (best possible sleep) to 10 (worst possible sleep).
Time Frame: Baseline (Day -7 to Day -1), Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
units on a scale | -1.0 (0.11) | -1.8 (0.11)

7. Secondary Outcome: Patient Reported Outcomes Measurement System (PROMIS) Fatigue
Description: Change from Baseline in the PROMIS score for fatigue at Week 12. The PROMIS fatigue short form 8a consists of 8 questions on a 5 point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40. Raw scores are converted to T-scores based on US population with score of 50 as average with a standard deviation of 10. Lower T-scores indicate less fatigue.
Time Frame: Day 1, Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
T-score | -4.2 (.47) | -6.4 (.47)

8. Secondary Outcome: Weekly Average of Daily Pain Diary
Description: Change from baseline to Week 12 in the weekly average of the daily self-reported average pain severity score using an 11-point (0-10) NRS. Scores range from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline (Day -7 to Day -1), Week 12
Population: Results are reported for the ITT population which includes all patients who were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
Number analyzed (Participants) | 257 | 262
units on a scale | -1.0 (0.11) | -1.5 (0.11)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: All data is reported for the Safety population, which is defined as all patients who were issued investigational product.
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 2.8 mg
All-Cause Mortality (participants affected / at risk) | 0/256 | 0/262
Serious Adverse Events (participants affected / at risk) | 4/256 | 3/262
Other Adverse Events (participants affected / at risk) | 17/256 | 132/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SL Tablet (N=256) | TNX-102 SL Tablet, 2.8 mg (N=262)
Seizure (Nervous system disorders) | 0 | 1 — Possible Seizure (unknown cause)
Pneumonia (Infections and infestations) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 — Near Syncopal Episode
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Non-cardiac Chest Pain (General disorders) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SL Tablet (N=256) | TNX-102 SL Tablet, 2.8 mg (N=262)
Hypoaesthesia Oral (Gastrointestinal disorders) | 2 | 105
Glossodynia (Gastrointestinal disorders) | 4 | 24
Paraesthesia Oral (Gastrointestinal disorders) | 3 | 20
Product Taste Abnormal (Product Issues) | 2 | 16
Fatigue (General disorders) | 6 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.